CLINICAL TRIAL: NCT04635111
Title: A Long-term Study to Further Evaluate the Risk of Hepatotoxicity Associated With TURALIO™ (Pexidartinib) Treatment
Brief Title: A Long-term Study Evaluating Hepatotoxicity Associated With TURALIO™ (Pexidartinib) Treatment
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: PL3397-A-U401
Record Dates: First submitted 2020-10-29; First posted 2020-11-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Hepatotoxicity; Tenosynovial Giant Cell Tumor
Keywords: Hepatotoxicity; Tenosynovial Giant Cell Tumor; Pexidartinib; TURALIO™
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath | interventions — pexidartinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The optional liver biopsy will be performed as soon as reasonably possible after the liver test abnormality criteria are first met and before liver tests have returned to normal. Four blood samples will be drawn on the day of, or up to 4 days before, the optional biopsy. One sample will evaluate liver test results (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP], gammaglutamyl transferase [GGT], total bilirubin [TBIL], direct bilirubin), serum creatinine, and blood urea nitrogen (BUN) at the study site. The remaining three samples will be used for central laboratory analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Symptomatic TGCT Participants: Adult patients with symptomatic TGCT associated with severe morbidity or functional limitations and not amenable to improvement with surgery, and who experience moderate or severe hepatotoxicity due to use of TURALIO™ (pexidartinib).
  Interventions: Drug: TURALIO™

INTERVENTIONS:
Drug: TURALIO™ — This is a non-interventional, observational study to evaluate long-term risk of hepatic failure associated with TURALIO™ (pexidartinib) treatment. No study medication will be provided to the participants.

SUMMARY:
A study to evaluate the long-term risk of hepatic failure with TURALIO™ (pexidartinib) and the mechanism of liver injury based upon optional liver biopsy information among patients who received or are receiving TURALIO™ (pexidartinib) and experience hepatotoxicity.

DETAILED DESCRIPTION:
This FDA post-marketing requirement study will evaluate the long-term risk of hepatic failure with TURALIO™ (pexidartinib) and the mechanism of liver injury based upon liver biopsy information among patients who received or are receiving TURALIO™ (pexidartinib) for symptomatic tenosynovial giant cell tumor (TGCT) associated with severe morbidity or functional limitations and not amenable to improvement with surgery, and who experience hepatotoxicity. An optional liver biopsy will be collected from enrolled patients for central laboratory analysis of macrophage and immune cell profiles to investigate possible mechanisms of the hepatotoxicity. Additionally, 4 blood samples will be collected to evaluate liver function, other relevant safety tests, peripheral immune cells, and for pharmacogenomic testing. Enrolled patients will be followed at least yearly for 10 years to assess long-term risk of hepatic failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with symptomatic TGCT associated with severe morbidity or functional limitations and not amenable to improvement with surgery
* Age ≥18 years old
* Emergence of at least one of the following liver test abnormalities due to TURALIO™ (pexidartinib) exposure:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 × upper limit of normal (ULN) with concurrent total bilirubin (TBIL) >2 × ULN
  * Isolated TBIL >2 × ULN (excluding patients with Gilbert's syndrome)
  * Isolated AST or ALT >10 × ULN
  * Alkaline phosphatase (ALP) >2 x ULN with gamma-glutamyl transferase (GGT) >2 x ULN
* Consent to study procedures, long-term safety follow-up, and use of data from the TURALIO™ (pexidartinib) Risk Evaluation and Mitigation Strategy (REMS) program

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with symptomatic TGCT associated with severe morbidity or functional limitations and not amenable to improvement with surgery, who experience moderate or severe hepatotoxicity due to TURALIO™ (pexidartinib).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2036-06-01 (Estimated); Study Completion 2036-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Hepatic Failure After Discontinuation of TURALIO™ (pexidartinib) | Baseline up to 10 years
  Hepatic failure is defined as severe liver injury with encephalopathy and impaired synthetic function (INR >= 1.5) as well as liver transplant and hepatic-related death.

SECONDARY OUTCOMES:
Number of Participants With Liver Test Abnormalities | Baseline up to 10 years
  Liver test abnormalities were defined as the following: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 × upper limit of normal (ULN) with concurrent total bilirubin (TBIL) >2 × ULN; Isolated TBIL >2 × ULN (excluding patients with Gilbert's syndrome); Isolated AST or ALT >10 × ULN; Alkaline phosphatase (ALP) >2 x ULN with gamma-glutamyl transferase (GGT) >2 x ULN.
Number of Participants With A Liver Transplant | Baseline up to 10 years
Number of Participants Experiencing Death | Baseline up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (8):
- United States (8):
  - Kamalesh K Sankhala MD INC, Santa Monica, California
  - Sarcoma Oncology Research Center LLC, Santa Monica, California
  - UCLA Hematology and Oncology, Santa Monica, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Montefiore Medical Center, New York, New York
  - OSU - James Comprehensive Cancer Center, Columbus, Ohio
  - Kelsey Seybold Clinic - Pearland, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/